CLINICAL TRIAL: NCT03456011
Title: Battlefield Acupuncture (BFA), an Adjunct Treatment During Sodium Hyaluronate Injections for Knee Osteoarthritis: A Prospective Pilot Study
Brief Title: Battlefield Acupuncture With Sodium Hyaluronate Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher Gomez, Orthopaedic PA Resident, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OrthoDSC
Record Dates: First submitted 2018-02-14; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFA with Eufflexa injections (Other): BFA treatment before Sodium Hyaluronate injections.
  Intervention: BFA
  Interventions: Other: Battlefield Acupuncture
- Anesthetic with Eufflexa injections (No Intervention): Receiving Standard of care determined by their provider
  No interventions

INTERVENTIONS:
Other: Battlefield Acupuncture — Battlefield Acupuncture gold semi permanent needles
  Arms: BFA with Eufflexa injections

SUMMARY:
The study evaluates pain relief and subsequent range of motion changes combining battlefield acupuncture with sodium hyaluronate vs local anesthetic and sodium hyaluronate

DETAILED DESCRIPTION:
Sodium hyaluronate is FDA approved for knee osteoarthritis. It is a widely used treatment for this condition. This does provide immediate pain relief and is often used in conjunction with lidocaine and ropivacaine to both improve pain relief and treatment tolerance.

battlefield acupuncture has been showing promise as an adjunct pain relief treatment option. If used during intra articular visco supplementation knee injections, this may provide pain relief and positive changes in range of motion without the need of local anesthetic being injected into the joint space.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the BAMC Orthopaedic clinic
* Active duty, dependent and civilians
* Ages 18-65
* Diagnosed with knee osteoarthritis by their Orthopaedic provider
* Determined to be eligible for Sodium Hyaluronate injections by their Orthopaedic provider

Exclusion Criteria:

* Patient without knee osteoarthritis diagnosis
* Patient requiring immediate surgery for their knee complaints
* Patients younger than 18 or older than 65
* Pregnant patients
* Patients without active pain
* Patients with history of knee arthroplasty
* Patients with auricular deformity which would affect BFA
* Patient with history of vasovagal secondary to needles or injections
* Patients with active infection at BFA treatment sites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 4 months
  Pain Scale. zero to 100 mm line. point on line if severity of pain. Zero no pain, 100 worst pain imaginable.

SECONDARY OUTCOMES:
Numerical Rating Scale | 4 months
  Pain Scale. Number pain scale 0-10. Zero no pain, 10 worst pain imaginable
KOOS | 4 months
  Knee function scoring. Questionnaire, scoring zero to 100. 100 is no pain or issues, zero is worst possible score.
KOOS Physical function short form | 4 months
  Knee function scoring. Questionnaire, scoring zero to 100. 100 is no pain or issues, zero is worst possible score.

CONTACTS AND LOCATIONS:
Locations (1):
- BAMC, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared within study group to include primary investigator and associate investigators. General demographic information will be collected to include in study results